CLINICAL TRIAL: NCT00698009
Title: Study to Infuse Haploidentical Natural Killer Cells in Patients With Relapsed or Refractory Neuroblastoma
Brief Title: Haploidentical Natural Killer (NK) Cells in Patients With Relapsed or Refractory Neuroblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0752
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Results first posted 2012-11-22 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Natural Killer Cell; NK Cell Infusion; Haploidentical Natural Killer (NK) Cells; Fludarabine; Fludarabine Phosphate; Fludara; Cyclophosphamide; Cytoxan; Neosar; Interleukin-2; IL-2; Proleukin; Mesna; Mesnex; Infusion of NK cells; Pediatric NK Cell Infusion; Pediatric Neuroblastoma; Pediatric NK; Pediatric
MeSH Terms: conditions — Neuroblastoma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Mesna; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fludarabine + Cyclophosphamide + NK Cell Infusion (Experimental): Fludarabine 25 mg/m^2 intravenous (IV) Daily Over 30 minutes Starting 6 days before the NK cell infusion (considered Day -6) and once a day through Day -2. Cyclophosphamide 60 mg/kg IV Daily Over 2 Hours On Days -5 and -4. Natural Killer Cell Infusion on Day 0. Mesna 12 mg/kg By Vein, Over about 15 minutes, 5 Times Per Day on Days -5 and -4. Interleukin-2 subcutaneously three times weekly for 9 total doses following NK Cell Infusion.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Natural Killer Cell Infusion; Drug: Mesna; Drug: Interleukin-2

INTERVENTIONS:
Drug: Fludarabine — 25 mg/m^2 By Vein Daily Over 30 minutes Starting 6 days before the NK cell infusion (considered Day -6) and once a day through Day -2.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Cyclophosphamide — 60 mg/kg By Vein Daily Over 2 Hours On Days -5 and -4
  Other Names: Cytoxan; Neosar
Biological: Natural Killer Cell Infusion — Natural Killer Cell Infusion on Day 0.
  Other Names: Infusion of NK cells; NK Cell Infusion
Drug: Mesna — 12 mg/kg By Vein, Over about 15 minutes, Five Times Per Day on Days -5 and -4.
  Other Names: Mesnex
Drug: Interleukin-2 — Received under skin three times weekly for 9 total doses following NK Cell Infusion:
  For patients weighing 45 kg or more, dose administered is 10 Million units three times weekly for 9 total doses. For patients less than 45 kg, dose administered is 5 Million units/m2 (max dose 10 Million units) three times weekly for 9 total doses.
  Other Names: IL-2; Proleukin

SUMMARY:
Primary:

Evaluate safety, feasibility, persistence, and anti-tumor effect of infused haploidentical donor-derived natural killer (NK) cells and low-dose interleukin-2 (IL-2).

Secondary:

* Quantification of cytokine levels;
* Assessment of NK cell immunophenotype and function.

DETAILED DESCRIPTION:
Experimental Therapy:

NK cells are part of the immune system (the cells in the body that naturally fight disease and infection). NK cells can sometimes destroy tumor cells, and they may be better at destroying tumor cells when the NK cells are "mismatched" for certain proteins called human leukocyte antigens (HLA). This can be determined by looking at the donor's and the recipient's HLA types and by checking for other specialized proteins on the donor's NK cells (called killer immunoglobulin receptors [KIR]).

The NK cells will be collected from the donor's blood and then processed using an experimental device called a CliniMACS device. This device is designed to separate out the NK cells from the rest of the donor's collected white blood cells, using a special magnet. Before being infused into the recipient (you, if you choose to take part), the collected NK cells will be treated with a study drug called interleukin-2 (IL-2) in order to try to activate the NK cells' killing ability. You will also receive IL-2 injections to try to help the NK cells survive after infusion and possibly increase in number.

Screening Tests:

Within 28 days before you can start treatment on this study, you will have "screening tests" to help the study doctor decide if you are eligible to take part in this study. The following tests will be performed:

* To check the status of the disease, you will have bone marrow aspirations and biopsies performed. To collect a bone marrow biopsy and aspirate, up to 2 areas of the hip bone are numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a needle.
* For another check of the status of the disease, you will most likely need to have computed tomography (CT) scans of the neck, sinuses, chest, stomach area (abdomen), and hip area (pelvis), and the brain.
* If the doctor thinks it is necessary, the status of the disease will also be checked with standard/routine tests such as positron emission tomography (PET) scans, iodine-131-meta- iodobenzylguanidine (MIBG -- a test that uses injected radioactive material and a special scanner to locate a tumor), and/or a bone scan.
* To measure your heart rate and level of oxygen in the blood, you will have a pulse oximetry test. This test uses a clothespin-shaped device that goes on the finger for about a minute.
* You will have a physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate).
* Your medical history will be recorded.
* Blood (about 4 tablespoons) will be drawn for routine tests and to check for diseases (infections such as the human immunodeficiency virus [HIV]). You will be told the results of this test for any diseases. If you have one of these infections, you will probably not be able to participate in this study.
* Urine or an additional 4 teaspoons of blood may also be drawn for other routine tests to check the disease status.
* Blood (up to 6 tablespoons) will be drawn and used to test for HLA and KIR typing, and you and the donor will be told the results of this test.
* Females who are able to have children must have a negative serum pregnancy test (as part of the blood sample described above, or possibly an additional 1 teaspoon).

These screening tests would also need to be repeated before an additional NK cell infusion for this study, in order to see if you continue to be eligible to receive one. This will be described further below.

Identifying an Eligible Donor:

Your relative, who must share half of your HLA genes to be eligible for the study, will be tested to see if his or her KIR molecule has the "mismatch" that researchers believe should help the donor's NK cells to target the tumor cells in your body.

The donor's blood will also be tested to guard against the possibility of transmitting an infection to you during the NK cell infusion.

Samples of the donor's blood will be used to help researchers develop future tests that will be used to track how long the infused NK cells survive and function in recipients' bodies. In order to help track the cells after infusion, researchers prefer (but do not require) that if you are a female recipient, your donor should be male and if you are a male recipient, your donor should be female.

Conditioning Phase:

If you are found to be eligible to take part in this study, you will start the "conditioning" phase of this study within 4 weeks after the screening tests. Over the course of 6 days, you will receive chemotherapy with cyclophosphamide and fludarabine to weaken your immune system in order to help the survival of the infused NK cells, and then mesna to protect your bladder from side effects that cyclophosphamide may cause.

Cyclophosphamide, fludarabine, and mesna will preferably be infused through an indwelling catheter (a tube that remains in a vein, such as tunneled in the arm or through the chest). If you already have an indwelling catheter in place, you will not need to have a new one placed. If a new catheter is needed, however, you will be asked to sign a separate informed consent form for its placement.

The Conditioning schedule is the following:

-Starting 6 days before the NK cell infusion (considered Day -6) and once a day through Day -2, you will receive fludarabine by vein, over about 30 minutes.

On Days -5 and -4, you will receive cyclophosphamide by vein, over about 2 hours each time.

-Five times per day on Days -5 and -4, you will receive mesna by vein, over about 15 minutes each time.

Infusion of NK Cells:

On Day 0 you will receive the NK cells by vein, preferably through an indwelling catheter. The doctor will decide what amount of NK cells will be infused, which will affect how long the infusion lasts, but usually it lasts less than 1 hour.

To help prevent an allergic reaction to the infused cells (such as fever and chills), you will receive Benadryl (diphenhydramine) by vein, over 15-30 minutes, and Tylenol (acetaminophen) by mouth. You will also receive fluids by vein to help decrease the risk of kidney damage.

You or a caregiver will be trained in how to perform the IL-2 injections yourself. This drug will be injected under the skin for 9 doses over the course of 3 weeks.

If the doctor decides you are not eligible to receive the NK cell infusion on Day 0, you will be taken off study without receiving the donor's NK cells. The collected NK cells will be thrown away.

Blood Test for Measuring NK Cell Survival:

Blood (up to 4 teaspoons each time) will be drawn and tested to see how long the NK cells survive in your body. This blood will be drawn on Day 0 (before the NK cell infusion and again 2 hours later) and on Days 2, 7, 14, 21, and 28. (It is possible that this blood draw schedule will stop earlier if the disease gets worse or the infused NK cells can no longer be seen.)

Possible Additional NK Cell Infusion:

If the neuroblastoma responds and you did not suffer a new intolerable side effect from the NK cells, then you may be eligible to receive 1 additional infusion of NK cells. If so, the rest of the study procedures would be the same as before (the screening tests to determine your eligibility, the requirement that the donor still be eligible, the Conditioning Phase with chemotherapy, the IL-2 injections, and the blood tests). You must use the same donor as before, if he or she is still eligible.

Hospitalization:

So that you can be monitored for side effects, you will need to stay in the hospital from Day -6 until after the NK cell infusion (or longer if medically necessary).

Follow-Up Visits:

After your final NK cell infusion, you will return for follow-up visits at least 3 times a week during the first 3 weeks. Then you will return for follow-up visits at around Day +28 and again 3 months after the last NK cell infusion. Following your 3 month visit, you will be asked to return for follow-up visits every 3 months up until one year after the last NK cell infusion. Below is a schedule of what will be done at each visit:

* Initial 3 weeks post infusion (3 times per week):
* Any changes in your medical history will be recorded, and a physical exam will be performed.
* Blood (up to 2 tablespoons) will be drawn for routine tests.

Day 28, at 3, 6, 9, and 12 months after infusion visits:

* Any changes in your medical history will be recorded, and a physical exam will be performed.
* Blood (up to 2 tablespoons) will be drawn for routine tests.
* Urine or an additional 4 teaspoons of blood may be drawn for other routine tests to check the disease status.
* CT scans of the neck, sinus, chest, abdomen, and pelvis will be performed, and a CT of the brain may also be performed if the study doctor feels it is needed.

MIBG scan may be performed if your tumor was positive on MIBG scan in the past or if your doctor feels it is needed.

-Bone marrow biopsies/aspirations may be performed once in the first month, then may be done at each visit if you had neuroblastoma in your bone marrow at the time you started on the study or if your doctor feels it is necessary.

PET scan and/or bone scan may be performed sometime in Months 2 or 3, and again in months 6 -12 if your doctor feels it is needed.

This is an investigational study. Cyclophosphamide, fludarabine, mesna, and IL-2 are commercially available but not FDA approved for use in neuroblastoma. Injecting IL-2 under the skin is not FDA approved for use in increasing the production of NK cells. The CliniMACS device is not commercially available or FDA approved. Infusing NK cells in patients with neuroblastoma is also considered experimental. At this time and for this purpose, NK cell infusions and the CliniMACS device are being used in research only.

Up to 10 recipients and 10 donors will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria: (Must be met within 28 days prior to initiating lymphodepleting conditioning regimen) The first two patients enrolled in this protocol, if they have undergone a previous autologous transplant, will need to be at least 6 months post-transplant and/or have available prior cryopreserved autologous peripheral blood stem cells. This criterion safeguards against the possibility that the lymphodepletion regimen may lead to prolonged myelosuppression in this patient population.
2. Evidence of relapse or progression of neuroblastoma after autologous peripheral blood stem-cell transplantation or similar aggressive therapy; high risk neuroblastoma that is refractory to standard induction therapy.
3. Measurable disease, with at least one of the following: One or more measurable radiographic abnormalities (X-ray, CT, MRI, PET); MIBG (metaiodobenzylguanidine) scan with uptake at a minimum of 1 site; Bone marrow with tumor cells seen on routine morphology (not by neuron specific enolase (NSE) staining or by immunocytology only). If the only bony or soft tissue lesion available for evaluation has been previously irradiated, the lesion must either a) have viable neuroblastoma on biopsy at least 4 weeks after radiation therapy or b) have measurable growth in the lesion after radiation.
4. Donor must be related to the recipient.
5. Off all systemic chemotherapeutic agents or retinoids for at least 21 days prior to NK infusion.
6. Platelets >/= 50,000 * 10^ 9/L and hemoglobin (Hgb) >/= 9 g/dL, unsupported by transfusions in last seven days.
7. absolute neutrophil count (ANC) >/= 1,000 * 10^ 9/L, unsupported by cytokines in last seven days.
8. Off prednisone or other immunosuppressive medications for at least 3 days prior to both the lymphodepleting regimen and the NK infusion (This excludes chronic low dose steroids for adrenal replacement which may be continued).
9. Karnofsky score or Lansky score >/= 60.
10. Adequate renal function defined as: Serum creatinine (Cr), for adults less than or equal to 2 mg/dL, for children less than or equal to 2 mg/dL or less than or equal to 2 times upper limit of normal (ULN) for age (whichever is less). If these criteria are not met, then recipient must have a Cr clearance greater than 60 mL/min/1.73m^2.
11. Adequate liver function defined as: Total bilirubin </=2 mg/dL and serum glutamate pyruvate transaminase (SGPT/Alanine aminotransferase, ALT) </= 2.5 * ULN for age (unless Gilbert's disease or abnormal liver function due to primary disease).
12. Pulmonary symptoms controlled by medication and pulse oximetry greater than or equal to 92% room air.
13. Females of childbearing potential (non childbearing is defined as premenarchal, greater than one year post-menopausal or surgically sterilized) must have a negative serum pregnancy test obtained within 2 weeks prior to registration and may not be breast feeding during the study. All males and females of childbearing potential are required to use a form of contraception considered effective and medically acceptable by the Investigator during the time of the study.
14. Donor must meet standard medical eligibility criteria for allogeneic stem cell donation and be able and willing to undergo apheresis.
15. Donor must have infectious disease marker testing [Hepatitis B, Hepatitis C, HIV, cytomegalovirus (CMV), Syphilis (RPR), Chagas, human T-cell lymphoma virus (HTLV), and West Nile Virus] and complete blood count (CBC), differential and platelet studies that meet standard medical eligibility criteria for allogeneic blood stem cell donation within 7 days of apheresis.
16. Donor, if a female of childbearing potential (non-childbearing is defined as premenarchal, greater than one year post-menopause or surgically sterilized), must have a negative serum pregnancy test obtained within 14 days of apheresis and may not be breast feeding.

Exclusion Criteria:

1. Exclusion Criteria: These criteria apply to both the start of the lymphodepleting regimen and to the NK infusion
2. Evidence of HIV (human immunodeficiency virus) disease or positive serology for HIV.
3. Currently requiring supplemental oxygen or on a ventilator.
4. Currently undergoing dialysis.
5. New detected cardiac arrhythmia not controlled with medical management within prior 72 hour period.
6. Hypotension requiring pressor support within prior 72 hour period.
7. Uncontrolled infection, daily fever greater than or equal to 39 degrees Celsius or new positive culture for bacteria, fungus, or virus within the 72 hours prior to NK-cell infusion.
8. Ascites requiring paracentesis within prior 72 hour period.
9. Seizure activity, clinically detectable encephalopathy or new focal neurologic deficits within prior 72 hour period.
10. Donor may not have an uncontrolled infection within 7 days of apheresis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan S. Kelly, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period June 05, 2008 to December 03, 2010. All recruitment done at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Fludarabine + Cyclophosphamide + NK Cell Infusion
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fludarabine + Cyclophosphamide + NK Cell Infusion
Number analyzed (Participants) | 1
Age, Continuous [Median (Standard Deviation); unit: years] | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Participant Disease Response
Description: Neuroblastoma International Response Criteria: Complete Response (CR): No evidence of disease (primary and metastasis) clinically & radiographic studies, (homovanillic acid (HVA)/vanillylmandelic acid (VMA) normal). Very Good Partial Response (VGPR): >90% reduction in primary tumor, resolution all metastatic tumor except bone. No new bone lesions and improvement on scan of all pre-existing lesions; HVA/VMA decreased >90%. Partial Response (PR): 50-90% reduction primary and all measurable metastatic lesions, 0-1 bone marrow samples with tumor; scans of bone lesions same as VGPR. HVA/VMA decreased 50-90%. Mixed Response (MR): > 50% reduction any measurable disease (primary or metastases); no new lesions; <25% increase in any existing lesion (exclude bone marrow evaluation). No Response (NR): No new lesions; < 25% increase in existing lesion. Progressive Disease (PD): Any new lesions. Increase <25% in measurable lesion, previous negative bone marrow positive for tumor.
Time Frame: 1 Year for overall patient response, or until disease progression
Arm/Group | Fludarabine + Cyclophosphamide + NK Cell Infusion
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants Infused Haploidentical Donor-derived Natural Killer (NK) Cells and Low-dose Interleukin-2 (IL-2)
Description: Feasibility of an infused allogeneic donor NK cell product and IL-2 following a cyclophosphamide and fludarabine preparative regimen to treat relapsed neuroblastoma after autologous peripheral blood stem cell (PBSC) transplant where feasibility is defined as being able to infuse NK cells on day 0.
Time Frame: 21 days, up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Fludarabine + Cyclophosphamide + NK Cell Infusion
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine + Cyclophosphamide + NK Cell Infusion (N=1)
Fever - Neutropenia (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No